CLINICAL TRIAL: NCT04687722
Title: Effects of High Intensity Aerobic Training on Primary Dysmenorrhea Among Young Females.
Brief Title: High Intensity Aerobic Training on Primary Dysmenorrhea
Acronym: HIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/00835 Iqra Imtiaz
Record Dates: First submitted 2020-12-25; First posted 2020-12-29 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Primary Dysmenorrhea
Keywords: pain; Dysmenorrhae symptoms; Menstrual Symptom Questionnaire
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated at the same time following their respective protocols.
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Aerobic Training Group. (Experimental): The experimental group will receive High Intensity Aerobic Training at 80-90% of Heart Rate Maximum calculated using karvonen rule.
  Interventions: Other: High Intensity Aerobic Training.
- Control Group (Active Comparator): The control group will receive routine low Intensity aerobic Training at 40-60% of Heart Rate Maximum calculated using karvonen rule.
  Interventions: Other: Low intensity Aerobic Training

INTERVENTIONS:
Other: High Intensity Aerobic Training. — Participants will perform 2-5 minutes of low to moderate intensity warm up exercises and then 20 minutes of high intensity aerobic training at 80-90% of heart rate maximum increased gradually on treadmill and elliptical trainer and then 2-5 minutes of low to moderate intensity cool down exercises.
  Arms: High Intensity Aerobic Training Group.
Other: Low intensity Aerobic Training — Participants will perform 2-5 minutes of low to moderate intensity warm up exercises and then 20 minutes of low intensity aerobic training at 40-60% of heart rate maximum increased gradually on elliptical trainer and jogging and then 2-5 minutes of low to moderate intensity cool down exercises.
  Arms: Control Group

SUMMARY:
Now a days Aerobic Exercise programs has been widely used as non-pharmacological means of treating pain disorders. This study intends to determine the effects of high intensity aerobic training on pain intensity, dysmenorrhea symptoms and quality of life of young girls having primary dysmenorrhea.

DETAILED DESCRIPTION:
This study is a Randomized Control Trial, which will be conducted in Shifa Tameer-e-Millat University (Department of Rehabilitation Sciences). the calculated Sample size is 24 individuals using Epitool with 95% Confidence Interval (CI) and power 80%. Individual will be screened out according to inclusion criteria. Individuals will be allocated randomly into two groups, 12 in High Intensity Aerobic training group and 12 in Low Intensity Aerobic Training group by sealed envelope method. High Intensity Aerobic Training will be use in experimental group. Low Intensity Aerobic Training will be used in Control group. Assessment will be done on baseline day 1 prior to the intervention and after 8 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried female students.
* Moderate to severe dysmenorrhea during the last three periods according to the Numeric Pain Rating Scale.

Exclusion Criteria:

* Presence of known chronic disease (heart disease, kidney, respiratory, asthma, diabetes, nervous disorders, blood pressure), limitation on sports/physical activities due to special medical problems.
* Presence of any disease of reproductive system.
* Irregular monthly cycle.
* Use of any particular medications affecting dysmenorrhea before or during the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants will be recruited in the study.
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline
  Numeric Pain Rating Scale (NPRS) will be used for measuring pain intensity of all participants by single examiner. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Numeric Pain Rating Scale (NPRS) | Post 8 weeks
  Numeric Pain Rating Scale (NPRS) will be used for measuring pain intensity of all participants by single examiner. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Menstrual Symptom Questionnaire | Baseline
  Menstrual Symptom Questionnaire will be used for measuring the severity of dysmenorrhea symptoms. It consisted of 25 items questions, participants are asked to indicate degree of their symptoms experience.
Menstrual Symptom Questionnaire | Post 8 weeks
  Menstrual Symptom Questionnaire will be used for measuring the severity of dysmenorrhea symptoms. It consisted of 25 items questions, participants are asked to indicate degree of their symptoms experience.

SECONDARY OUTCOMES:
SF-36 questionnaire | Baseline
  SF-36 questionnaire will be used for assessing the quality of life of all participants.
SF-36 questionnaire | Post 8 weeks
  SF-36 questionnaire will be used for assessing the quality of life of all participants.
Serum Progesteron level | Baseline
  Blood samples will be taken to measure Serum Progesteron level
Serum Progesteron level | Post 8 weeks
  Blood samples will be taken to measure Serum Progesteron level

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Shifa Tameer-e-Millat University (Department of Rehabilitation Sciences)., Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaziri F, Hoseini A, Kamali F, Abdali K, Hadianfard M, Sayadi M. Comparing the effects of aerobic and stretching exercises on the intensity of primary dysmenorrhea in the students of universities of bushehr. J Family Reprod Health. 2015 Mar;9(1):23-8. PMID 25904964
- [Background] Ortiz MI, Cortes-Marquez SK, Romero-Quezada LC, Murguia-Canovas G, Jaramillo-Diaz AP. Effect of a physiotherapy program in women with primary dysmenorrhea. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:24-9. doi: 10.1016/j.ejogrb.2015.08.008. Epub 2015 Aug 17. PMID 26319652
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Kannan P, Claydon LS, Miller D, Chapple CM. Vigorous exercises in the management of primary dysmenorrhea: a feasibility study. Disabil Rehabil. 2015;37(15):1334-9. doi: 10.3109/09638288.2014.962108. Epub 2014 Sep 22. PMID 25243766
- [Background] Dehnavi ZM, Jafarnejad F, Kamali Z. The Effect of aerobic exercise on primary dysmenorrhea: A clinical trial study. J Educ Health Promot. 2018 Jan 10;7:3. doi: 10.4103/jehp.jehp_79_17. eCollection 2018. PMID 29417063